CLINICAL TRIAL: NCT03726411
Title: The Effect of Non-surgical Periodontal Therapy on the Gingival Crevicular Fluid Levels of Prolactin Hormone in Patients With Periodontitis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eman Mohamed Amr (Other)
Responsible Party: Sponsor-Investigator, Eman Mohamed Amr, Associate Professor of Oral Medicine and Periodontology, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Prolactin 101
Record Dates: First submitted 2018-10-30; First posted 2018-10-31 (Actual); Last update posted 2019-03-12 (Actual); Status verified 2019-03

CONDITIONS: Periodontitis; Prolactin in GCF
Keywords: periodontitis; Prolactin; GCF; non-surgical periodontal treatment
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- periodontitis group (Experimental): in this group, prolactin in GCF will be assessed at baseline and after 3 months of receiving non-surgical periodontal treatment
  Interventions: Procedure: non-surgical periodontal therapy
- control group (No Intervention): in this group of systemically and periodontally healthy participants, prolactin in GCF will be assessed at baseline only

INTERVENTIONS:
Procedure: non-surgical periodontal therapy — scaling and root planing
  Arms: periodontitis group

SUMMARY:
The present study will be conducted on fifty participants. All participants will receive a full-mouth clinical examination, and the following periodontal parameters will be recorded: Plaque Index (PI). Gingival Index (GI), probing depth (PD), and clinical attachment level (CAL). All of these measurements will be recorded at six sites at baseline for all participants and 3 months after non-surgical periodontal therapy for the study group. GCF samples will be collected from the buccal aspects of teeth that had the highest signs of inflammation and attachment loss for periodontitis group at baseline and 3 months after non-surgical periodontal therapy. As for controls, the samples will be collected from buccal aspect of upper first molar at baseline. The samples will be assayed for prolactin by using an enzyme linked immunosorbent assay kits (Elisa) according to the manufacturer instruction.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with moderate to severe chronic periodontitis, with probing pocket depth (PPD) ≥ 4-6 mm and clinical attachment level ≥ 4-5 mm, according to the American Academy of Periodontology.7
* Highly motivated and cooperative patients

Exclusion Criteria:

* The presence of any systemic disease.
* Taking medications for the last 3 months before conducting this study.
* Pregnancy and lactation.
* Any type of previous periodontal treatment (surgical or non-surgical) in the preceding 6 months.
* Smoking (former or current).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
prolactin in GCF | 3 months
  prolactin level in GCF by ELISA

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided